CLINICAL TRIAL: NCT00023556
Title: Genetic Architecture of Heart Disease in Rural Brazil
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 982; R01HL066480-05 (NIH)
Record Dates: First submitted 2001-09-07; First posted 2001-09-07 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-08

CONDITIONS: Chagas Disease; Heart Diseases; Arrhythmia; Heart Failure, Congestive
MeSH Terms: conditions — Chagas Disease; Heart Diseases; Arrhythmias, Cardiac; Heart Failure

SUMMARY:
To examine the genetics of human susceptibility to Chagas' disease, a leading cause of heart disease throughout Latin America.

DETAILED DESCRIPTION:
BACKGROUND:

Chagas' disease is a leading cause of heart disease throughout Latin America, affecting between 16 and 18 million individuals. The disease, named after the Brazilian physician Carlos Chagas who first described it in 1909, exists only on the American Continents. It is caused by a flagellate protozoan parasite, Trypanosoma cruzi, transmitted to humans by blood-sucking triatomine insects known popularly in the different countries as "vinchuca", "barbeiro", "chipo" etc. The geographical distribution of the human T.cruzi infection extends from Mexico to the south of Argentina. In Brazil alone, approximately 10 percent of the population is seropositive for T. cruzi. Given the large pool of primary hosts for this zoonotic disease, complete eradication of Chagas' disease through control of the arthropod vector is unlikely. Research with humans and animal models indicates that there is variation in susceptibility to infection, and disease outcome, and that this variation may be due to genetic factors. Thus, this form of heart disease represents a complex phenotype with potential genetic determinants to both susceptibility to infection and differential disease pathogenesis.

DESIGN NARRATIVE:

The genetic epidemiology project studies an estimated 1,125 Black individuals age 18 years or older from a small community in Posse, Brazil in which the study population may be drawn from as few as four to five large pedigrees with varying blood relationships. Preliminary pilot data appear very promising regarding the primary hypothesis that specific genetic factors influence the susceptibility to this complex zoonotic disease. The investigation will be divided into three parts involving phenotypic characterization, statistical genetic analyses to determine the relative proportion of the phenotypic variance due to additive genetic effects, and localization of genes influencing the development of Chagas' disease.

The phenotypic characterization will involve clinical history, infection status, immunologic studies, and cardiac status. The chronic phase of T. cruzi infection results in Chagas' disease manifest as a cardiomyopathy with heart block, conduction disturbance, ventricular tachyarrhythmia, heart failure, and sudden arrhythmic death. The cardiac phenotyping will involve electrocardiographic time intervals (PR interval, QRS duration, QT interval duration) as well as abnormal patterns (left anterior fascicular block, left ventricular hypertrophy, right bundle branch block), and possibly some measure of heart failure in terms of New York Heart Association functional classification. Right bundle branch block is probably the most frequent early manifestation of chronic cardiac involvement.

The genetic linkage studies will attempt to localize genes influencing susceptibility to T. cruzi infection, ECG parameters (e.g., right bundle branch block), and immunologic factors using markers placed approximately every 10 centimorgans (cM) throughout the genome.

About 375 individuals will be sampled per year. Each subject will donate two 10 ml samples of blood which will be used for immunoassays for seropositivity for T. cruzi, and for genotyping with 382 polymorphic short tandem repeats. During the initial visits, the population subjects will also be interviewed to gather information on demographic, pedigree, and socioeconomic makeup. Additionally, questions on pregnancy status, household ecology (years in the house, rooms shared, pets, rodents, food storage, triatomid bug history, etc) and residence history will be determined during the survey. In the fourth year, the investigators will return to the collection site and administer ECGs on 375 individuals per year.

The blood collected in Brazil will be sent to San Antonio for high-throughput genotyping using 382 polymorphic short tandem repeats (STRs) spread throughout the genome. A population specific 10cM map is expected to be useful for linkage analysis.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Williams-Blangero — Southwest Foundation for Biomedical Research

REFERENCES:
- [Background] Williams-Blangero S, VandeBerg JL, Blangero J, Correa-Oliveira R. Genetic epidemiology of Trypanosoma cruzi infection and Chagas' disease. Front Biosci. 2003 May 1;8:e337-45. doi: 10.2741/1058. PMID 12700060